CLINICAL TRIAL: NCT06276738
Title: The LINFU® U.S. Registry for the Detection of Pancreatic Ductal Adenocarcinoma (PDAC) in Patients With Clinical Signs and/or Symptoms of Disease
Brief Title: The LINFU® U.S. Registry in Patients With Clinical Signs and/or Symptoms of Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Adenocyte, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Adenocyte 102
Record Dates: First submitted 2024-02-18; First posted 2024-02-26 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Pancreatic Cancer; Jaundice; Abdominal Neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms; Jaundice; Abdominal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Slides and cell blocks made from pancreatic fluid collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients at increased risk for developing pancreatic cancer: Patients who exhibit symptoms suggestive of PDAC (i.e. jaundice, abdominal pain, weight loss, nausea and vomiting etc.) or have evidence of imaging studies suggestive of PDAC will undergo LINFU® testing.
  Interventions: Diagnostic Test: LINFU® (Low Intensity Non-Focused Ultrasound excitation of the pancreas)

INTERVENTIONS:
Diagnostic Test: LINFU® (Low Intensity Non-Focused Ultrasound excitation of the pancreas) — Patients will undergo low intensity non-focused ultrasound excitation of the pancreas for a total of 15 minutes. A contrast agent will be administered IV at five minute intervals. The patient will then receive a dose of secretin and the the patient's pancreatic juice will then be collected for a total of 15 minutes.

SUMMARY:
Evaluate LINFU® in patients who exhibit signs or symptoms (i.e. jaundice, abdominal pain, weight loss, nausea and vomiting etc.) suggestive of pancreatic cancer (PDAC) or have evidence of imaging studies suggestive of PDAC.

DETAILED DESCRIPTION:
Adenocyte has developed a proprietary pancreatic cancer detection method, LINFU®, (Low Intensity Non-Focused Ultrasound excitation of the pancreas) that increases the sensitivity of pancreatic juice cytology. LINFU® excitation of circulating microbubbles increases the exfoliation of pancreatic ductal cells. The sensitivity of cytological examination of the pancreatic fluid obtained by LINFU® can also be potentially enhanced by neural network-based computer-assisted analysis.

In this study, LINFU® will be evaluated in patients who exhibit symptoms suggestive of PDAC (i.e. jaundice, abdominal pain, weight loss, nausea and vomiting etc.) or have evidence of imaging studies suggestive of PDAC. In addition, patients with PDAC identified only with LINFU® and not detected with other diagnostic tests will be followed long term to determine the progression rate of these tumors and to determine whether LINFU® results in earlier intervention, treatment and improvement in patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Both males and females will be enrolled and must be at least 18 years of age and under age of 90
* Patients, who in the opinion of the Investigator, require biopsy to rule out PDAC because they display at least one of the following or both: a) clinical symptoms of PDAC including jaundice, nausea and vomiting, weight loss, abdominal pain, bloating or the feeling of fullness, itchy skin, lower back pain, light-colored, greasy stools, sudden onset type 2 diabetes, etc. b) one or more imaging studies suggestive of PDAC
* All patients must undergo contemporaneous imaging, either within 90 days before the LINFU® procedure or within 30 days after the procedure, with one or more of the following: EUS± FNA, MRI/MRCP, ERCP, CT or CEUS.
* Institutional Review Board (IRB)-approved consent must be signed by patients to participate in this study.

Exclusion Criteria:

* Patient under the age of 18 and over the age 90
* Contraindications to LINFU®/EUS/ERCP as determined by study investigators: Patient with uncorrectable coagulopathy; Patient that cannot undergo anesthesia due to cardiopulmonary contraindication as deemed by the anesthesiologist; Unstable medically (cardiopulmonary, neurologic, or cardiovascular status)
* Patients undergoing EUS or ERCP for a suspected bile duct cancer arising from the intrahepatic or extrahepatic biliary epithelium
* Patients who are already known to have PDAC by cytologic or histologic evidence
* Patients with intraductal papillary mucinous neoplasm of the pancreas (IPMN) identified either before the study or during the study through imaging evaluation will be excluded
* Pregnant females will be excluded
* Patient that is unable to provide informed consent
* Patient with known allergy to the microbubble contrast agent or secretin

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: High risk patients with either clinical symptoms or imaging abnormalities or both, being evaluated for PDAC.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2034-03-01 (Estimated); Study Completion 2034-05-01 (Estimated)

PRIMARY OUTCOMES:
The number of pancreatic ductal adenocarcinomas identified only with LINFU® will be compared to standard screening methods | 5 years
  The total number of pancreatic ductal adenocarcinomas identified with LINFU® by analysis of pancreatic fluid will be compared to the number of these lesions identified with current screening tests, including endoscopic ultrasound ± fine needle aspiration (EUS± FNA),magnetic resonance imaging / magnetic resonance cholangiopancreatography (MRI/MRCP), endoscopic retrograde cholangiopancreatography (ERCP),computed tomography (CT) or contrast-enhanced ultrasound (CEUS).

SECONDARY OUTCOMES:
The change in size of pancreatic ductal adenocarcinomas identified only with LINFU® will be determined | 5 years
  Patients with pancreatic ductal adenocarcinomas identified only with LINFU® and not detected with other diagnostic tests will be monitored long- term (5 years) by EUS- FNA, MRI/MRCP, ERCP, CT and CEUS to assess whether these tumors increase in size (measured in mm) and to determine how many require medical or surgical intervention.
Determine the number of patients with pancreatic ductal adenocarcinoma identified only with LINFU® that require medical or surgical intervention | 5 years
  Patients with pancreatic ductal adenocarcinomas identified only with LINFU® and not detected with other diagnostic tests will be monitored long- term (5 years) by EUS- FNA, MRI/MRCP, ERCP, CT and CEUS to assess whether these tumors increase and how many require medical or surgical intervention.

OTHER OUTCOMES:
Yearly survival rate of patients with pancreatic ductal adenocarcinomas identified only with LINFU® | 5 years
  Patients will be followed by EUS- FNA, MRI/MRCP, ERCP, CT and CEUS and yearly survival rates of patients with pancreatic ductal adenocarcinomas identified only with LINFU® and not detected with other diagnostic tests will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Haber, Principal Investigator — Manhattan Endoscopy Center

IPD SHARING:
Plan to Share IPD: No